CLINICAL TRIAL: NCT05209646
Title: Bee Honey as a Therapeutic Modality for Children With Functional Dyspepsia
Brief Title: Bee Honey and Functional Dyspepsia in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, mamdouh abdulmaksoud abdulrhman, Professor of Pediatrics, Ain Shams University, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MS 513/ 2021
Record Dates: First submitted 2021-12-11; First posted 2022-01-26 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Functional Gastrointestinal Disorders
Keywords: Functional dyspepsia in children; Bee honey
MeSH Terms: conditions — Gastrointestinal Diseases | interventions — pteropsin, Apis mellifera

STUDY DESIGN:
Intervention Model Description: Two groups; interventional and control groups
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trial (Intervention) group (Experimental): Patients will receive honey for 8 weeks in a dose of 30 ml undiluted honey per day divided as 5 ml honey 30 minutes before each meal six times daily. The honey will be kept in a closed glass container and away from light until the time of use. Each patient will be provided with a well-sealed container containing 210 ml honey each week. The honey used in the study will be a raw, unprocessed Clover honey collected from AL Mahala-Gharbia governorate, Egypt. The honey will be supplied directly from a beekeeper without heating or gamma irradiation
  Interventions: Dietary Supplement: Bee honey
- Control (Non-intervention) group (No Intervention): No honey will be given to this group

INTERVENTIONS:
Dietary Supplement: Bee honey — patients will receive honey for 8 weeks in a dose of 30 ml undiluted honey per day divided as 5 ml honey 30 minutes before each meal six times daily. The honey will be kept in a closed glass container and away from light until the time of use. Each patient will be provided with a well-sealed container containing 210 ml honey each week. The honey used in the study will be a raw, unprocessed Clover honey collected from AL Mahala-Gharbia governorate, Egypt. The honey will be supplied directly from a beekeeper without heating or gamma irradiation.
  Arms: Trial (Intervention) group

SUMMARY:
Functional dyspepsia is a constellation of diverse gastrointestinal disturbing symptoms with multifactorial feature, varying from upper abdominal bloating to nausea and vomiting, that are not attributable to organic causes after proper medical assessment. Treatment options are unsatisfactory due to the lack of identifiable pathophysiology as well as the pharmacological therapy are less effective, so using an additional reliable non-pharmacological therapy would be promising.

Bee honey has not only being used as food but also it has being used as an alternative medicine for its several benefits in different health aspects. This study will address the use of bee honey as an adjuvant therapy to functional dyspepsia in children under proper follow-up periods.

DETAILED DESCRIPTION:
Functional dyspepsia (FD), among the most common gastrointestinal (GIT) disorders, is characterized by early satiation, postprandial fullness, epigastric pain, or epigastric burning in the absence of an organic or metabolic disease. FD is not a life-threatening serious illness, but its symptoms could persist; rather, they limit one's social life and reduce their quality of life. In addition, FD constitutes a serious disease burden worldwide because of its high prevalence.

Proton pump inhibitor (PPI) in the form of Omeprazole had the best result on all dyspeptic symptoms being relieved on children aged 3-18 years with dyspepsia.

Nonetheless, the efficacy of pharmacological therapies remains unsatisfactory and a considerable number of FD patients are refractory to conventional pharmacological treatments. Furthermore, low compliance of the traditional therapy can be observed in some FD patients as they would opt out from these pharmacological options because of the concerns on the side effects. In the absence of an approved drug to treat FD many patients seek person-centered, nonpharmacological approaches.

As the consumption of nutrients can moderate the sensors of the upper gastrointestinal tract movement, changes in diet can probably improve the symptoms of functional dyspepsia. Alternative and complementary medicine has also been proposed as a practical treatment for dyspepsia. Another substance used for treating this disorder is honey, which is economical and has a short treatment period. Many old sources have reported the use of honey for preventing stomach ulcers, gastritis, and gastroenteritis. Honey has a stimulating effect on the stomach nerves, which may be due to the antioxidant activity of honey. According to a study, the consumption of honey reduces the acidic activity of the stomach by 56%. Another study showed the effect of honey on the improved blood supply of stomach microscopic capillaries and it helped in the repair of ulcers. The symptoms of functional dyspepsia can also be improved through diet education. In various studies, most people have reported the onset or exacerbation of dyspepsia symptoms after eating. Unhealthy nutritional behaviors can exacerbate the symptoms of functional dyspepsia.

Adjuvant supplementation of honey based formulation of Nigella sativa can cause significant symptomatic improvement of patients with functional dyspepsia.

Honey is considered one of the most common foods having alleviating effects on non-ulcer dyspepsia.

In considerations of scarce knowledge in this field, health attributes of bee honey as a reliable therapy to improve the symptoms of functional dyspepsia in children, deserves seeking for.

ELIGIBILITY:
Inclusion Criteria:

* All patients between 8 and 18 years-old, based on Rome IV criteria that provide evidence-based definitions and classifications for so-called functional gastrointestinal disorders, such as functional dyspepsia in children and adolescents, with 1 or more of the following bothersome symptoms at least 4 days per month for at least 2 months:
* Postprandial fullness
* Early satiation
* Epigastric pain or burning not associated with defecation
* After appropriate evaluation, the symptoms cannot be fully explained by another medical condition
* Postprandial distress syndrome includes bothersome postprandial fullness or early satiation that prevents finishing a regular meal. Supportive features include upper abdominal bloating, postprandial nausea, or excessive belching.
* Epigastric pain syndrome, which includes all of the following: bothersome (severe enough to interfere with normal activities) pain or burning localized to the epigastrium. The pain is not generalized or localized to other abdominal or chest regions and is not relieved by defecation or passage of flatus. Supportive criteria can include (a) burning quality of the pain but without a retrosternal component and (b) the pain commonly induced or relieved by ingestion of a meal but may occur while fasting.

Exclusion Criteria:

* The presence of alarm symptoms and signs which might suggest underlying organic pathology as listed in Rome III criteria including: (Persistent right upper or right lower quadrant pain, dysphagia, persistent vomiting, gastrointestinal blood loss, nocturnal diarrhea, family history of inflammatory bowel disease, celiac disease, or peptic ulcer disease, pain that wakes the child from sleep, arthritis, perirectal disease, involuntary weight loss, deceleration of linear growth, delayed puberty or unexplained fever).
* Gastrointestinal tract surgery, one year post-operative.
* Diabetes mellitus
* Any debilitating disorder e.g. malignancy, severe malnutrition, renal failure, etc.
* Patients on medications that may produce GIT disorders e.g. aspirin, steroids or NSAIDs

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2022-01-21 (Actual); Primary Completion 2022-06-21 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Effect of bee honey on functional dyspepsia as an adjuvant therapy among dyspepsia suffering children assessed by Modified Glasgow Dyspepsia Severity Score in comparison to age and sex matched controls. | 6 months
  * Every week during the first 4 weeks of the study. Patients' response will be divided into complete recovery, partial improvement, no improvement or worsening of symptoms. At the 4th week of the study, those who completely recovered or partially improved will discontinue using PPI, while those with no improvement or worsening will continue on PPI and will be excluded
  * At the 8th week of the study, honey will be discontinued and reassessment will be done
  * Assessment of the severity of dyspepsia using "Modified Glasgow Dyspepsia Severity Score". It will be tried to evaluate the frequency of abdominal pain (predominant symptom), the number of school or preschool days of absenteeism, the duration and intensity of pain, the presence of nocturnal pain and vomiting. Scores ranged from 0 to16, with high scores indicating greater severity. According to this scale patients will be divided with dyspepsia into three groups: Mild (score <6), moderate (score 7-10) and severe (score >11)

SECONDARY OUTCOMES:
Effect of bee honey on recurrence of symptoms one month after stopping medications assessed by Modified Glasgow Dyspepsia Severity Score. | 6 months
  * Assessment of patients will be done at the 12th week of the study, patients in both groups will be reassessed and any recurrence of symptoms in the complete recovery patients or flare up of symptoms among those with partial recovery will be documented.
  * Assessment of the severity of dyspepsia using "Modified Glasgow Dyspepsia Severity Score". It will be tried to evaluate the frequency of abdominal pain (predominant symptom), the number of school or preschool days of absenteeism, the duration and intensity of pain, the presence of nocturnal pain and vomiting. Scores ranged from 0 to16, with high scores indicating greater severity. According to this scale patients will be divided with dyspepsia into three groups: Mild (score <6), moderate (score 7-10) and severe (score >11)

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akhondi-Meybodi M, Aghaei MA, Hashemian Z. The role of diet in the management of non-ulcer dyspepsia. Middle East J Dig Dis. 2015 Jan;7(1):19-24. PMID 25628849
- [Background] Dehghani SM, Imanieh MH, Oboodi R, Haghighat M. The comparative study of the effectiveness of cimetidine, ranitidine, famotidine, and omeprazole in treatment of children with dyspepsia. ISRN Pediatr. 2011;2011:219287. doi: 10.5402/2011/219287. Epub 2011 Apr 5. PMID 22389770
- [Background] Febriani TB, Widowati T and Juffrie M Reducing dyspeptic symptoms in children: proton pump inhibitor vs. H2 receptor antagonist. Paediatrica Indonesiana. 2014; 54(4):198-201.
- [Background] Hyams JS, Di Lorenzo C, Saps M, Shulman RJ, Staiano A and Van Tilburg M. Childhood functional gastrointestinal disorders: child/adolescent. Gastroenterology. 2016; 150(6):1456-1468. e2.
- [Background] Kim YS, Kim N. Functional Dyspepsia: A Narrative Review With a Focus on Sex-Gender Differences. J Neurogastroenterol Motil. 2020 Jul 30;26(3):322-334. doi: 10.5056/jnm20026. PMID 32606255
- [Background] Koppen IJ, Nurko S, Saps M, Di Lorenzo C, Benninga MA. The pediatric Rome IV criteria: what's new? Expert Rev Gastroenterol Hepatol. 2017 Mar;11(3):193-201. doi: 10.1080/17474124.2017.1282820. Epub 2017 Jan 24. PMID 28092724
- [Background] Mohtashami R, Huseini HF, Heydari M, Amini M, Sadeqhi Z, Ghaznavi H, Mehrzadi S. Efficacy and safety of honey based formulation of Nigella sativa seed oil in functional dyspepsia: A double blind randomized controlled clinical trial. J Ethnopharmacol. 2015 Dec 4;175:147-52. doi: 10.1016/j.jep.2015.09.022. Epub 2015 Sep 18. PMID 26386381
- [Background] Pesce M, Cargiolli M, Cassarano S, Polese B, De Conno B, Aurino L, Mancino N, Sarnelli G. Diet and functional dyspepsia: Clinical correlates and therapeutic perspectives. World J Gastroenterol. 2020 Feb 7;26(5):456-465. doi: 10.3748/wjg.v26.i5.456. PMID 32089623
- [Background] Rasquin A, Di Lorenzo C, Forbes D, Guiraldes E, Hyams JS, Staiano A, Walker LS. Childhood functional gastrointestinal disorders: child/adolescent. Gastroenterology. 2006 Apr;130(5):1527-37. doi: 10.1053/j.gastro.2005.08.063. PMID 16678566
- [Background] Samarghandian S, Farkhondeh T, Samini F. Honey and Health: A Review of Recent Clinical Research. Pharmacognosy Res. 2017 Apr-Jun;9(2):121-127. doi: 10.4103/0974-8490.204647. PMID 28539734
- [Background] Spiroglou K, Paroutoglou G, Nikolaides N, Xinias I, Giouleme O, Arsos G et al. Dyspepsia in childhood. Clinical manifestations and management. Annals of Gastroenterology. 2004; 17(2):173-180.
- [Background] Taghvaei T, Bagheri-Nesami M and Nikkhah A. The Effect of Honey and Diet Education on Symptoms of Functional Dyspepsia: A Randomized Clinical Trial. Iranian Red Crescent Medical Journal. 2018; 20(8): e65557.
- [Background] Wang YP, Herndon CC, Lu CL. Non-pharmacological Approach in the Management of Functional Dyspepsia. J Neurogastroenterol Motil. 2020 Jan 30;26(1):6-15. doi: 10.5056/jnm19005. PMID 31751504
- [Background] Yagi M, Homma S, Kubota M, Iinuma Y, Kanada S, Kinoshita Y, Ohtaki M, Yamazaki S, Murata H. The herbal medicine Rikkunshi-to stimulates and coordinates the gastric myoelectric activity in post-operative dyspeptic children after gastrointestinal surgery. Pediatr Surg Int. 2004 Jan;19(12):760-5. doi: 10.1007/s00383-003-1053-y. Epub 2004 Jan 9. PMID 14714134
- See also: Related Info — https://doi.org/10.14238/pi54.4.2014.198-201
- See also: Related Info — https://doi.org/10.1053/j.gastro.2016.02.015
- See also: Related Info — http://www.annalsgastro.gr/index.php/annalsgastro/article/view/288
- See also: Related Info — https://www.sid.ir/FileServer/JE/88120180806.pdf